CLINICAL TRIAL: NCT01885559
Title: HALT Progression of Polycystic Kidney Disease Study B
Acronym: HALT PKD B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Boehringer Ingelheim (Industry); Merck Sharp & Dohme LLC (Industry); Polycystic Kidney Disease Foundation (Other); University of Pittsburgh (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HALT PKD B; U01DK062401 (NIH); U01DK082230 (NIH); NCT00067977 (obsolete NCT alias)
Record Dates: First submitted 2013-06-17; First posted 2013-06-25 (Estimated); Results first posted 2015-03-10 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Kidney, Polycystic
Keywords: polycystic kidney disease; polycystic; kidney; disease; adpkd; halt; pkd; blood pressure; bp; hypertension; renal; renin-angiotensin-aldosterone-system; RAAS
MeSH Terms: conditions — Polycystic Kidney Diseases; Disease; Polycystic Kidney, Autosomal Dominant; Familial paroxysmal dystonia; Hypertension | interventions — Lisinopril; Angiotensin-Converting Enzyme Inhibitors; Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ACE-I + placebo (Placebo Comparator): Monotherapy of lisinopril and placebo. Standard blood pressure control of 110-130/80 mm Hg
  Interventions: Drug: Lisinopril; Drug: Placebo
- ACE-I + ARB (Active Comparator): Dual therapy of lisinopril and telmisartan treatments. Standard blood pressure control of 110-130/80 mm Hg.
  Interventions: Drug: Lisinopril; Drug: Telmisartan

INTERVENTIONS:
Drug: Lisinopril — Lisinopril titrated to 5mg, 10mg, 20mg, 40mg as tolerated by participants, to achieve standard blood pressure control of 110-130/80 mm Hg.
  Other Names: ACE-I; ACE; Ace-Inhibitor
Drug: Telmisartan — Telmisartan titrated to 40mg and 80mg, as tolerated by participants, to achieve standard blood pressure control of 110-130/80 mm Hg.
  Other Names: ARB
  Arms: ACE-I + ARB
Drug: Placebo — Placebo titrated to 40mg and 80mg, as tolerated by participants, to achieve standard blood pressure control of 110-130/80 mm Hg.
  Other Names: Control
  Arms: ACE-I + placebo

SUMMARY:
The efficacy of interruption of the renin-angiotensin-aldosterone system (RAAS) on the progression of cystic disease and on the decline in renal function in autosomal dominant kidney disease (ADPKD) will be assessed in two simultaneous multicenter randomized clinical trials targeting different levels of kidney function: 1) early disease defined by GFR >60 mL/min/1.73 m2 (Study A); and 2) moderately advanced disease defined by GFR 25-60 mL/min/1.73 m2 (Study B). Participants will be recruited and enrolled, either to Study A or B, over the first three years. Participants enrolled in Study B will be followed for five-to-eight years, with the average length of follow-up being six and a half years.

Combination therapy will use angiotensin-converting-enzyme inhibitor (ACE-I) and an angiotensin-receptor blocker (ARB). Monotherapy will use ACE-I alone.

DETAILED DESCRIPTION:
* Specific Aim of Study B

To study the effects of ACE-I/ARB combination therapy as compared to ACE-I monotherapy in the setting of standard blood pressure control (110-130/80 mm Hg) on the time to a 50% reduction of baseline estimated Glomerular Filtration Rate (eGFR), end-state renal disease (ESRD) or death, in hypertensive individuals with moderate renal insufficiency (GFR 25-60 mL/min/1.73m2).

* Hypothesis to be tested in Study B

In hypertensive ADPKD individuals with moderate renal insufficiency (GFR 25-60 mL/min/1.73 m2), intensive blockade of the RAAS using combination ACE-I/ARB therapy will slow the decline in kidney function over ACE-I monotherapy, independent of standard blood pressure control (110-130/80 mm Hg).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADPKD.
* Age 15-49 (Study A); Age 18-64 (Study B).
* GFR >60 mL/min/1.73 m2 (Study A); GFR 25-60 mL/min/1.73 m2 (Study B).
* BP ≥130/80 or receiving treatment for hypertension.
* Informed Consent.

Exclusion Criteria:

* Pregnant/intention to become pregnant in 4-6 yrs.
* Documented renal vascular disease.
* Spot urine albumin-to-creatinine ratio of >0.5 (Study A) or ≥1.0 (Study B) and/or findings suggestive of kidney disease other than ADPKD.
* Diabetes requiring insulin or oral hypoglycemic agents / fasting serum glucose of >126 mg/dl / random non-fasting glucose of >200 mg/dl.
* Serum potassium >5.5 milliequivalent (mEq) /L for participants currently on ACE-I or ARB; >5.0 mEq/L for participants not currently on ACE-I or ARB.
* History of angioneurotic edema or other absolute contraindication for ACE-I or ARB. Intolerable cough associated with ACE-I is defined as a cough developing within six months of initiation of ACE-I in the absence of other causes and resolving upon discontinuation of the ACE-I.
* Indication (other than hypertension) for β-blocker or calcium channel blocker therapy (e.g. angina, past myocardial infarction, arrhythmia), unless approved by the site principal investigator. (PI may choose to accept an individual who is on only a small dose of one of these agents and would otherwise be eligible.)
* Systemic illness necessitating nonsteroidal antiinflammatory drugs (NSAIDs), immunosuppressant or immunomodulatory medications.
* Systemic illness with renal involvement.
* Hospitalized for acute illness in past 2 months.
* Life expectancy <2 years.
* History of non-compliance.
* Unclipped cerebral aneurysm >7mm diameter.
* Creatine supplements within 3 months of screening visit.
* Congenital absence of a kidney (also total nephrectomy for Study B).
* Known allergy to sorbitol or sodium polystyrene sulfonate.
* Exclusions specific to magnetic resonance (MR) imaging (Study A).

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 486 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schrier, M.D., Study Chair — University of Colorado, Denver; Arlene Chapman, M.D., Principal Investigator — Emory University; Ronald Perrone, M.D., Principal Investigator — Tufts University-New England Medical Center; Vicente Torres, M.D., Principal Investigator — Mayo Clinic; Marva Moxey-Mims, M.D., Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Charity G Moore, PhD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tufts University-New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository, https://repository.niddk.nih.gov/studies/halt-pkd/?query=halt%20pkd
URL: https://repository.niddk.nih.gov/studies/halt-pkd/?query=halt%20pkd

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Chebib FT, Zhou X, Garbinsky D, Davenport E, Nunna S, Oberdhan D, Fernandes A. Tolvaptan and Kidney Function Decline in Older Individuals With Autosomal Dominant Polycystic Kidney Disease: A Pooled Analysis of Randomized Clinical Trials and Observational Studies. Kidney Med. 2023 Apr 14;5(6):100639. doi: 10.1016/j.xkme.2023.100639. eCollection 2023 Jun. PMID 37250503
- [Derived] Torres VE, Abebe KZ, Chapman AB, Schrier RW, Braun WE, Steinman TI, Winklhofer FT, Brosnahan G, Czarnecki PG, Hogan MC, Miskulin DC, Rahbari-Oskoui FF, Grantham JJ, Harris PC, Flessner MF, Moore CG, Perrone RD; HALT-PKD Trial Investigators. Angiotensin blockade in late autosomal dominant polycystic kidney disease. N Engl J Med. 2014 Dec 11;371(24):2267-76. doi: 10.1056/NEJMoa1402686. Epub 2014 Nov 15. PMID 25399731
- See also: Polycystic Kidney Disease Foundation Website — http://www.pkdcure.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for HALT PKD Study B occurred at seven clinical sites between February 2006 and June 2009.
Groups:
- ACE-I + Placebo: ACE-I + placebo and standard blood pressure control of 110-130/80 mm Hg
  Lisinopril and Placebo: Lisinopril titrated to 5mg, 10mg, 20mg, 40mg and placebo titrated to 40mg and 80mg, as tolerated by participants, to achieve standard blood pressure control of 110-130/80 mm Hg.
- ACE-I + Angiotensin Receptor Blocker (ARB): ACE-I + angiotensin receptor blocker (ARB) and standard blood pressure control of 110-130/80 mm Hg
  Lisinopril and Telmisartan: Lisinopril titrated to 5mg, 10mg, 20mg, 40mg and telmisartan titrated to 40mg and 80mg, as tolerated by participants, to achieve standard blood pressure control of 110-130/80 mm Hg.
Period: Overall Study
Arm/Group | ACE-I + Placebo | ACE-I + Angiotensin Receptor Blocker (ARB)
Started | 242 | 244
Completed | 218 | 208
Not Completed | 24 | 36
Not completed — Lost to Follow-up | 15 | 16
Not completed — Less than full participation | 9 | 19
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ACE-I + ARB: ACE-I + ARB and standard blood pressure control of 110-130/80 mm Hg
  Lisinopril and Telmisartan: Lisinopril titrated to 5mg, 10mg, 20mg, 40mg and telmisartan titrated to 40mg and 80mg, as tolerated by participants, to achieve standard blood pressure control of 110-130/80 mm Hg.
- Total: Total of all reporting groups
Arm/Group | ACE-I + Placebo | ACE-I + ARB | Total
Number analyzed (Participants) | 242 | 244 | 486
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (8.1) | 48.6 (8.5) | 48.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 129 | 251
  Male | 120 | 115 | 235
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 224 | 230 | 454
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 0 | 1 | 1
PKD Genotype [Number; unit: participants]
  PKD1 | 183 | 179 | 362
  PKD2 | 30 | 30 | 60
  No Mutation Detected | 11 | 14 | 25
  No data | 18 | 21 | 39
Age at Diagnosis of Autosomal Dominant Polycystic Kidney Disease (yrs) [Mean (Standard Deviation); unit: years] | 33.5 (12.4) | 33.0 (12.0) | 33.2 (12.2)
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 28.0 (5.5) | 28.0 (4.9) | 28.0 (5.2)
Serum Creatinine (mg/dl) [Mean (Standard Deviation); unit: mg/dl] | 1.6 (0.4) | 1.5 (0.4) | 1.6 (0.4)
Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) eGFR (ml/min/m^2) [Mean (Standard Deviation); unit: ml/min/m^2] | 47.9 (12.2) | 48.5 (11.5) | 48.2 (11.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 50% Reduction of Baseline eGFR, End Stage Renal Disease (ESRD, Initiation of Dialysis or Preemptive Transplant), or Death.
Time Frame: Patients followed for 5-8 years with average of 6.5 years follow up
Population: Intention to Treat analysis was used for the primary outcome
Measure: Number; unit: participants
Arm/Group | ACE-I + Placebo | ACE-I + ARB
Number analyzed (Participants) | 242 | 243
participants | 116 | 115
Statistical Analysis 1: Comparison: ACE-I + Placebo vs ACE-I + ARB; Test type: Superiority or Other; p = 0.58, Regression, Cox; Analyses were adjusted for age, sex, race, baseline estimated Glomerular Filtration Rate (eGFR) and clinical site; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.82 to 1.42] — ACE+ARB (Lisinopril-telmisartan) compared to ACE+placebo (Lisinopril-placebo)

2. Secondary Outcome: Albuminuria
Description: Annual percent change in 24 hour urine albumin, centrally processed. Data from multiple years were analyzed with the primary focus on the change over time for the measure (from the slope of the model). The measure presented is the average annual percent change across the 8 years.
Time Frame: up to 8 years (annually assessed)
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: annual percent change
Arm/Group | ACE-I + Placebo | ACE-I + ARB
Number analyzed (Participants) | 242 | 243
annual percent change | 7.5 [5.2 to 9.9] | 7.3 [4.9 to 9.7]
Statistical Analysis 1: Comparison: ACE-I + Placebo vs ACE-I + ARB; Test type: Superiority or Other; p = 0.88, shared parameter model; shared parameter models used due to informative censoring that occurred when patients did not have secondary outcomes measured after reaching endpoint; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-3.2 to 2.8]

3. Secondary Outcome: Aldosterone
Description: Annual percent change in urinary aldosterone, centrally processed measure. Data from multiple years were analyzed with the primary focus on the change over time for the measure (from the slope for time from the model). The measure presented is the average annual percent change across the 8 years.
Time Frame: up at 8 years (annually assessed)
Population: Intention to treat analyses
Measure: Mean (95% Confidence Interval); unit: annual percent change
Arm/Group | ACE-I + Placebo | ACE-I + ARB
Number analyzed (Participants) | 242 | 243
annual percent change | -8.8 [-10.5 to -7.2] | -10.2 [-11.9 to -8.6]
Statistical Analysis 1: Comparison: ACE-I + Placebo vs ACE-I + ARB; Test type: Superiority or Other; p = 0.17, Mixed Models Analysis — controlling for age, sex, race, and clinical site; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-3.9 to 0.7] — ACE-I+ARB annual percent change minus ACE-I + placebo annual percent change

4. Secondary Outcome: Hospitalizations
Description: Hospitalization for any cause
Time Frame: up to 8 years
Population: Intention to treat analysis
Measure: Number; unit: events
Arm/Group | ACE-I + Placebo | ACE-I + ARB
Number analyzed (Participants) | 242 | 243
events | 173 | 136
Statistical Analysis 1: Comparison: ACE-I + Placebo vs ACE-I + ARB; Test type: Superiority or Other; p = 0.85, Regression, Cox; adjusting for age, sex, race, and clinical site and recurrent events; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.80 to 1.32] — Hazard ratio compares ACE-I + ARB compared to ACE-I + placebo

5. Secondary Outcome: Cardiovascular Hospitalizations
Description: Cause-specific hospitalizations (cardiovascular)
Time Frame: up to 8 years
Population: Intention to Treat analysis
Measure: Number; unit: events
Arm/Group | ACE-I + Placebo | ACE-I + ARB
Number analyzed (Participants) | 242 | 243
events | 29 | 16
Statistical Analysis 1: Comparison: ACE-I + Placebo vs ACE-I + ARB; Test type: Superiority or Other; p = 0.57, Regression, Cox; adjusting for age, sex, race, and clinical site and accounting for recurrent events; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.42 to 1.6] — Hazard ratio is comparing ACE-I + ARB to ACE-I + placebo

6. Secondary Outcome: Quality of Life Physical Component Summary
Description: Short Form-36 Quality of Life Physical Component Summary ranges from 0 (worst possible outcome) to 100 (best possible outcome). Data from multiple years were analyzed with the primary focus on the change over time for the measure (from the slope for time from the model). The measure presented is the average annual change across the 8 years.
Time Frame: up to 8 years (annually assessed)
Population: Intention to Treat analysis
Measure: Mean (95% Confidence Interval); unit: units on a scale per year
Arm/Group | ACE-I + Placebo | ACE-I + ARB
Number analyzed (Participants) | 242 | 243
units on a scale per year | -0.64 [-0.79 to -0.50] | -0.68 [-0.84 to -0.52]
Statistical Analysis 1: Comparison: ACE-I + Placebo vs ACE-I + ARB; Test type: Superiority or Other; p = 0.75, shared parameter model; Shared parameter models were used due to informed censoring when patients who reached the primary endpoint were no longer assessed on the measure; Mean Difference (Final Values) = -0.032, 95% CI 2-sided [-0.23 to 0.16]

7. Secondary Outcome: Quality of Life Mental Component Summary
Description: Short Form-36 Quality of Life Mental Component Summary ranges from 0 (worst possible outcome) to 100 (best possible outcome). Data from multiple years were analyzed with the primary focus on the change over time for the measure (from the slope for time from the model). The measure presented is the average annual change across the 8 years.
Time Frame: up to 8 years (annually assessed)
Population: Intention to treat analysis
Measure: Mean (95% Confidence Interval); unit: units on a scale per year
Arm/Group | ACE-I + Placebo | ACE-I + ARB
Number analyzed (Participants) | 242 | 243
units on a scale per year | -0.031 [-0.19 to 0.12] | -0.079 [-0.24 to 0.08]
Statistical Analysis 1: Comparison: ACE-I + Placebo vs ACE-I + ARB; Test type: Superiority or Other; p = 0.66, shared parameter model; Shared parameter models were used due to the informative censoring when patients who reached endpoint were not longer assessed on this measure; Mean Difference (Final Values) = -0.047, 95% CI 2-sided [-0.26 to 0.16]

8. Secondary Outcome: Back or Flank Pain
Description: Report of back or flank pain since the last visit (yes or no)
Time Frame: 48 months
Population: Cross sectional analysis at 48 months is reported only for those participants responding at that time point. Intention to treat analysis was used for in the modeling over time to incorporate all repeated measures.
Measure: Number (95% Confidence Interval); unit: percentage of participants at 48 months
Arm/Group | ACE-I + Placebo | ACE-I + ARB
Number analyzed (Participants) | 184 | 179
percentage of participants at 48 months | 43 [36 to 50] | 46 [39 to 53]
Statistical Analysis 1: Comparison: ACE-I + Placebo vs ACE-I + ARB; Test type: Superiority or Other; p = 0.64, Mixed Models Analysis; Generalized linear mixed models are used with a logit link. Model controlled for baseline age, sex, race, and clinical site; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.99 to 1.01] — Odds ratio represents the multiplicative effect of ACE-I + ARB group compared to the ACE-I + placebo group in change in pain over time. ACE-I + ARB OR per month was 1.01 (1.00, 1.01) and ACE-I + placebo OR was 1.01 (1.01, 1.01)

ADVERSE EVENTS:
Time Frame: Serious adverse event data were collected during follow up between 5-8 years with average follow up time of 5.2 years.
Arm/Group | ACE-I + Placebo | ACE-I + ARB
Serious Adverse Events (participants affected / at risk) | 88/242 | 88/244
Other Adverse Events (participants affected / at risk) | 66/242 | 60/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACE-I + Placebo (N=242) | ACE-I + ARB (N=244)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial infarction (Cardiac disorders) | 6 (6) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (2) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 15 (16) | 2 (5)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 6 (7) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 3 (4) | 1 (2)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 6 (6) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (2) | 3 (3)
Kidney infection (Infections and infestations) | 2 (2) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Injury to carotid artery (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bladder anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 7 (7)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Pregnancy, puerperium and perinatal conditions - Other, specify (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 1 (2)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 9 (11) | 4 (4)
Renal calculi (Renal and urinary disorders) | 2 (5) | 1 (1)
Renal colic (Renal and urinary disorders) | 4 (7) | 0 (0)
Renal hemorrhage (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (3) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 3 (3)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 12 (12) | 15 (21)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (5) | 3 (3)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACE-I + Placebo (N=242) | ACE-I + ARB (N=244)
Acute Kidney Injury (Renal and urinary disorders) | 32 (51) | 22 (31)
Hyperkalemia (Metabolism and nutrition disorders) | 41 (65) | 46 (70)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No